CLINICAL TRIAL: NCT03671473
Title: Comparison of Focused and Radial Extracorporeal Shock Wave for Carpal Tunnel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It is difficult to enroll patients
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB: 1-107-05-074
Record Dates: First submitted 2018-07-31; First posted 2018-09-14 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Extracorporeal shock wave
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused (Experimental): fESWT (0.05-0.29 mJ/mm2, 2000 shocks, 5 Hz)
  Interventions: Device: Extracorporeal shock wave
- Radial (Active Comparator): rESWT (2000shocks, 4 Bar, 5Hz)
  Interventions: Device: Extracorporeal shock wave

INTERVENTIONS:
Device: Extracorporeal shock wave — Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs). Different studies and clinical experiments have demonstrated the efficacy of shock waves in the treatment of musculoskeletal system such as chronic tendinopathies or hypertrophic pseudoarthrosis.

SUMMARY:
Extracorporeal shock wave is a novel treatment for peripheral nerve entrapment. This study was designed to compare the efficacy of focused and radial extracorporeal shock wave for carpal tunnel syndrome.

DETAILED DESCRIPTION:
Both focused and radial extracorporeal shock wave had been proved to treat carpal tunnel syndrome by several studies. However, there was no study comparing these two methods. Considering different mechanisms and costs, this randomized comparative trial would be conducted to compare the efficacy of focused and radial extracorporeal shock wave for carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and electrophysiological diagnosis of CTS

Exclusion Criteria:

* Cervical radiculopathy
* Polyneuropathy
* Brachial plexopathy
* Thoracic outlet syndrome
* Previous wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) at 24th weeks after treatment | Change of the mean of total SSS and FSS from baseline at 24th weeks after treatment
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of carpal tunnel syndrome which encompasses two components. eleven questions and eight items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Each question or item ranges from 1 to 5 with a higher score indicating severer symptom or a higher degree of disability. Total score of SSS ranges from 11-55 and FSS from 8-40. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | Pre-treatment, 2nd, 4th, 8th, 12th and 24th weeks after treatment
  Digital pain severity or paresthesia/dysthesia within 1 week prior to evaluation was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Nerve conduction velocity | Pre-treatment, 2nd, 4th, 8th, 12th and 24th weeks after treatment
  Change from baseline in conduction velocity of median nerve on 2nd, 4th, 8th,12th and 24th weeks after treatment.
Cross-sectional area (CSA) of the median nerve | Pre-treatment, 2nd, 4th, 8th, 12th and 24th weeks after treatment
  Change from baseline in cross-sectional area of the median nerve on 2nd, 4th, 8th, 12th and 24th weeks after treatment.
Nerve conduction amplitude | Pre-treatment, 2nd, 4th, 8th, 12th and 24th weeks after treatment
  Change from baseline in conduction amplitude of median nerve on 2nd, 4th, 8th,12th and 24th weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

REFERENCES:
- [Result] Wu YT, Ke MJ, Chou YC, Chang CY, Lin CY, Li TY, Shih FM, Chen LC. Effect of radial shock wave therapy for carpal tunnel syndrome: A prospective randomized, double-blind, placebo-controlled trial. J Orthop Res. 2016 Jun;34(6):977-84. doi: 10.1002/jor.23113. Epub 2015 Dec 10. PMID 26610183
- [Result] Ke MJ, Chen LC, Chou YC, Li TY, Chu HY, Tsai CK, Wu YT. The dose-dependent efficiency of radial shock wave therapy for patients with carpal tunnel syndrome: a prospective, randomized, single-blind, placebo-controlled trial. Sci Rep. 2016 Dec 2;6:38344. doi: 10.1038/srep38344. PMID 27910920
- [Result] Paoloni M, Tavernese E, Cacchio A, D'orazi V, Ioppolo F, Fini M, Santilli V, Mangone M. Extracorporeal shock wave therapy and ultrasound therapy improve pain and function in patients with carpal tunnel syndrome. A randomized controlled trial. Eur J Phys Rehabil Med. 2015 Oct;51(5):521-8. Epub 2015 Feb 20. PMID 25697763